CLINICAL TRIAL: NCT03228680
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre Trial Assessing the Efficacy and Safety of FE 999049 in Controlled Ovarian Stimulation in Japanese Women Undergoing an Assisted Reproductive Technology Programme
Brief Title: Efficacy and Safety of FE 999049 in Controlled Ovarian Stimulation in Japanese Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000273
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2021-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin delta; FE 999049; follitropin beta

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follitropin delta (Experimental): FE 999049 was administered as single daily subcutaneous injections in the abdomen. Participants randomized to FE 999049 had their individual dose determined on the basis of their anti-Müllerian hormone (AMH) level at screening and their body weight at randomization. The daily FE 999049 dose was fixed throughout the stimulation period. The minimum allowed daily FE 999049 dose was 6 μg and maximum allowed daily dose was 12 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
  Interventions: Drug: Follitropin delta
- Follitropin beta (Active Comparator): FOLLISTIM was administered as single daily subcutaneous injections in the abdomen. The starting dose of FOLLISTIM was 150 IU and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 375 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
  Interventions: Drug: Follitropin beta

INTERVENTIONS:
Drug: Follitropin delta — Single daily subcutaneous administration through pre-filled injection pen
  Other Names: FE 999049; REKOVELLE
  Arms: Follitropin delta
Drug: Follitropin beta — Single daily subcutaneous injection in the abdomen
  Other Names: FOLLISTIM
  Arms: Follitropin beta

SUMMARY:
To demonstrate non-inferiority of FE 999049 compared to FOLLISTIM with respect to number of oocytes retrieved in Japanese IVF/ICSI patients undergoing controlled ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Documents signed prior to any trial-related procedures.
* In good physical and mental health.
* Japanese females between the ages of 20 and 40 years.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II (defined by the revised American Society for Reproductive Medicine (ASRM) classification) or with partners diagnosed with male factor infertility, eligible for in vitro fertilization (IVF) and/or intracytoplasmic sperm injection (ICSI) treatment using ejaculated sperm from male partner.
* Infertility for at least 1 year before randomization (not applicable in case of tubal or severe male factor infertility).
* The trial cycle will be the participant's first controlled ovarian stimulation cycle for IVF/ICSI.
* Hysterosalpingography, hysteroscopy, saline infusion sonography or transvaginal ultrasound documenting a uterus consistent with expected normal function (e.g. no evidence of clinically interfering uterine fibroids defined as submucous or intramural fibroids larger than 3 cm in diameter, no polyps and no congenital structural abnormalities which are associated with a reduced chance of pregnancy) within 1 year prior to screening. This also includes women who have been diagnosed with any of the above medical conditions but have had them surgically corrected within 1 year prior to screening.
* Transvaginal ultrasound documenting presence and adequate visualization of both ovaries, without evidence of significant abnormality (e.g. no endometrioma greater than 3 cm or enlarged ovaries which would contraindicate the use of gonadotropins) and fallopian tubes and surrounding tissue without evidence of significant abnormality (e.g. no hydrosalpinx) within 1 year prior to screening. Both ovaries must be accessible for oocyte retrieval.
* Early follicular phase (cycle day 2-4) serum levels of follicle stimulating hormone (FSH) between 1 and 15 IU/L (results obtained within 3 months prior to screening).
* Body mass index (BMI) between 17.5 and 32.0 kg/m^2 (both inclusive) at screening.

Exclusion Criteria:

* Known endometriosis stage III-IV (defined by the revised ASRM classification).
* One or more follicles >10 mm (including cysts) observed on the transvaginal ultrasound prior to start of stimulation on stimulation day 1 (puncture of cysts prior randomization is allowed).
* Known history of recurrent miscarriage (defined as three consecutive losses after ultrasound confirmation of pregnancy (excl. ectopic pregnancy) and before week 24 of pregnancy).
* Known abnormal karyotype of participant or of her partner. In case the sperm production is severely impaired (concentration <1 million/mL), normal karyotype, including no Y chromosome microdeletion, must be documented.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Any known clinically significant systemic disease (e.g. insulin-dependent diabetes).
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the trial with the exception of controlled thyroid function disease.
* Known tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotropins.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 373 (Actual)
Dates: Start 2017-07-29 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (17):
- Japan (17):
  - Yachiyo Hospital, Anjo, Aichi-ken
  - Investigational Site 8121, Chiba, Chiba
  - Yokota Maternity Hospital, Maebashi, Gunma
  - Sophia Ladies Clinic, Sagamihara, Kanagawa
  - Investigational Site 8122, Sendai, Miyagi
  - Investigational Site 8123, Higashiōsaka-shi, Osaka
  - Investigational Site 8120, Osaka, Osaka
  - Ladies Clinic Kitahama, Osaka, Osaka
  - Investigational Site 8125, Saitama-shi, Saitama
  - Investigational Site 8124, Shinjuku-Ku, Tokyo
  - Akita University Hospital, Akita
  - Yamashita Ladies' Clinic, Hyōgo
  - Investigational Site 8126, Saitama
  - Omiya Ladies Clinic, Saitama
  - Saint Women's Clinic, Saitama
  - Women's Clinic Fujimino, Saitama
  - Tokushima University Hospital, Tokushima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ishihara O, Arce JC; Japanese Follitropin Delta Phase 3 Trial (STORK) Group. Individualized follitropin delta dosing reduces OHSS risk in Japanese IVF/ICSI patients: a randomized controlled trial. Reprod Biomed Online. 2021 May;42(5):909-918. doi: 10.1016/j.rbmo.2021.01.023. Epub 2021 Feb 9. PMID 33722477
- [Result] Ishihara O, Nelson SM, Arce JC. Comparison of ovarian response to follitropin delta in Japanese and White IVF/ICSI patients. Reprod Biomed Online. 2022 Jan;44(1):177-184. doi: 10.1016/j.rbmo.2021.09.014. Epub 2021 Sep 23. PMID 34799275
- [Result] Fernandez-Sanchez M, Fatemi H, Garcia-Velasco JA, Heiser PW, Daftary GS, Mannaerts B. Incidence and severity of ovarian hyperstimulation syndrome (OHSS) in high responders after gonadotropin-releasing hormone (GnRH) agonist trigger in "freeze-all" approach. Gynecol Endocrinol. 2023 Dec;39(1):2205952. doi: 10.1080/09513590.2023.2205952. PMID 37156263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 investigational sites in Japan randomized participants to the trial between 29 July 2017 to 08 July 2019.
Pre-assignment Details: A total of 373 participants were screened. Of these, 25 were screening failures and 348 participants were randomized: 170 participants were exposed to FE 999049 & 177 participants were exposed to FOLLISTIM. One participant was randomized to FOLLISTIM but not exposed to investigational medicinal product (IMP) was considered a randomization failure.
Groups:
- FE 999049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen. Participants randomized to FE 999049 had their individual dose determined on the basis of their anti-Müllerian hormone (AMH) level at screening and their body weight at randomization. The daily FE 999049 dose was fixed throughout the stimulation period. The minimum allowed daily FE 999049 dose was 6 μg and maximum allowed daily dose was 12 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- FOLLISTIM (Follitropin Beta): FOLLISTIM was administered as single daily subcutaneous injections in the abdomen. The starting dose of FOLLISTIM was 150 IU and fixed for the first five stimulation days, after which it could be adjusted by 75 IU based on the individual response. The maximum allowed daily dose was 375 IU. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
Period: Overall Study
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Started | 170 | 178
Completed | 147 | 143
Not Completed | 23 | 35
Not completed — Adverse Event | 13 | 18
Not completed — Randomization failure | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- FE 999049 (Follitropin Delta): FE 999049 was administered as single daily subcutaneous injections in the abdomen. Participants randomized to FE 999049 had their individual dose determined on the basis of their AMH level at screening and their body weight at randomization. The daily FE 999049 dose was fixed throughout the stimulation period. The minimum allowed daily FE 999049 dose was 6 μg and maximum allowed daily dose was 12 μg. Dosing continued until the criterion for triggering of final follicular maturation was met. Participants could be treated for a maximum of 20 days.
- Total: Total of all reporting groups
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta) | Total
Number analyzed (Participants) | 170 | 177 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] — Number analyzed differs from the overall population as one participant in the FOLLISTIM (Follitropin beta) group was randomized but not exposed to treatment.
  years | 34.2 (3.5) | 34.0 (3.4) | 34.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Number analyzed differs from the overall population as one participant in the FOLLISTIM (Follitropin beta) group was randomized but not exposed to treatment.
  Participants
    Female | 170 | 177 | 347
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number analyzed differs from the overall population as one participant in the FOLLISTIM (Follitropin beta) group was randomized but not exposed to treatment.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 170 | 177 | 347
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number analyzed differs from the overall population as one participant in the FOLLISTIM (Follitropin beta) group was randomized but not exposed to treatment.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 170 | 177 | 347
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Number analyzed differs from the overall population as one participant in the FOLLISTIM (Follitropin beta) group was randomized but not exposed to treatment.
  participants
    Japan | 170 | 177 | 347

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: 36h (± 2h) after triggering of final follicular maturation (On day of oocyte retrieval)
Population: The full analysis set (FAS) comprised all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: Oocytes retrieved
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Oocytes retrieved | 9.3 (5.4) | 10.5 (6.1)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Mean number of oocytes retrieved; Test type: Non-Inferiority — The pre-specified non-inferiority (NI) margin was -3.0 oocytes. The NI was evaluated based on the two-sided 95% CI from the ANOVA on 'number of oocytes retrieved' with treatment and AMH stratum as fixed factors; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.3 to -0.1] — If the lower bound of 95% CI was well above pre-specified NI limit of -3.0 oocytes, then NI of FE 999049 to FOLLISTIM with respect to number of oocytes retrieved in women undergoing controlled ovarian stimulation would be demonstrated

2. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical pregnancy was defined as at least one gestational sac 5-6 weeks after transfer.
Time Frame: 5-6 weeks after transfer (up to approximately 3 months after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants | 25.3 | 23.7
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Percentage of participants with at least one gestational sac 5-6 weeks after transfer; Test type: Other; Risk Difference (RD) = 1.6, 95% CI 2-sided [-7.5 to 10.6] — The difference (FE 999049-FOLLISTIM) in rates was estimated and a two-sided 95% Cl was constructed using the Mantel-Haenszel method to combine results across AMH strata

3. Secondary Outcome: Positive Beta Unit of Human Chorionic Gonadotropin (Beta-hCG) Rate
Description: Defined as positive serum beta-hCG test 13-15 days after transfer.
Time Frame: 13-15 days after transfer (up to approximately 1.5 months after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants | 29.4 | 29.4
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Percentage of participants with positive beta-hCG; Test type: Other; Risk Difference (RD) = 0.0, 95% CI 2-sided [-9.5 to 9.6] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Vital Pregnancy Rate
Description: Vital pregnancy was defined as at least one intrauterine gestational sac with fetal heart beat 5-6 weeks after transfer.
Time Frame: 5-6 weeks after transfer (up to approximately 3 months after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants | 23.5 | 21.5
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Percentage of participants with vital pregnancy; Test type: Other; Risk Difference (RD) = 2.0, 95% CI 2-sided [-6.7 to 10.8] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Implantation Rate
Description: Implantation rate was defined as the number of gestational sacs 5-6 weeks after transfer divided by the number of blastocysts transferred.
Time Frame: 5-6 weeks after transfer (up to approximately 3 months after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants with blastocyst transfer.
Measure: Number; unit: % of sacs/blastocysts transferred
Units Other Than Participants: Embryos transferred
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Number analyzed (Embryos transferred) | 135 | 141
% of sacs/blastocysts transferred | 31.9 | 29.8
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Percentage of implanted embryos 5-6 weeks after transfer; Test type: Other; Risk Difference (RD) = 1.9, 95% CI 2-sided [-8.9 to 12.8] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Proportion of Participants With Cycle Cancellation Due to Poor or Excessive Ovarian Response
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants
  Cycle cancelled due to poor ovarian response | 1.2 | 0.6
  Cycle cancelled due to excessive ovarian response | 0 | 1.1

7. Secondary Outcome: Proportion of Participants With Blastocyst Transfer Cancellation Due to Excessive Ovarian Response / OHSS Risk
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants | 7.6 | 11.3
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with blastocyst transfer cancellation; Test type: Superiority; p = 0.244, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors

8. Secondary Outcome: Proportion of Participants With <4, 4-7, 8-14, 15-19 and ≥20 Oocytes Retrieved
Description: Defined as proportion of participants grouped according to the number of oocytes retrieved. The proportion of participants with <4 oocytes (low response), 4-7 oocytes (moderate response), 8-14 oocytes (targeted response), 15-19 oocytes (hyperresponse) and ≥20 oocytes (severe hyperresponse) are presented.
Time Frame: On the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 173
percentage of participants
  Low response (<4 oocytes) | 8.3 | 5.2
  Moderate response (4-7 oocytes) | 36.1 | 26.6
  Targeted response (8-14 oocytes) | 40.8 | 42.8
  Hyperresponse (15-19 oocytes) | 10.1 | 14.5
  Severe hyperresponse (≥ 20 oocytes) | 4.7 | 11.0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with <4 oocytes retrieved (low response); Test type: Superiority; p = 0.254, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with 4-7 oocytes retrieved (moderate response); Test type: Superiority; p = 0.041, Regression, Logistic — P-value was based on likelihood ratio test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 3: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with 8-14 oocytes retrieved (targeted response); Test type: Superiority; p = 0.705, Regression, Logistic — P-value was based on likelihood ratio test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 4: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with 15-19 oocytes retrieved (hyperresponse); Test type: Superiority; p = 0.183, Regression, Logistic — P-value was based on likelihood ratio test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 5: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with >= (more than equal to) 20 oocytes retrieved (severe hyperresponse); Test type: Superiority; p = 0.030, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors

9. Secondary Outcome: Proportion of Participants With Extreme Ovarian Responses (Defined as <4, ≥15 or ≥20 Oocytes Retrieved) in Risk Population
Time Frame: On the day of oocyte retrieval (up to 22 days after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 173
percentage of participants
  AMH < 15 pmol/L (<4 oocytes retrieved): number analyzed (Participants) | 69 | 73
  AMH < 15 pmol/L (<4 oocytes retrieved) | 11.6 | 12.3
  AMH >= 15 pmol/L (>=15 oocytes retrieved): number analyzed (Participants) | 100 | 100
  AMH >= 15 pmol/L (>=15 oocytes retrieved) | 22.0 | 42.0
  AMH >= 15 pmol/L (>=20 oocytes retrieved): number analyzed (Participants) | 100 | 100
  AMH >= 15 pmol/L (>=20 oocytes retrieved) | 8.0 | 19.0
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with extreme ovarian responses: AMH < 15 pmol/L (<4 oocytes retrieved); Test type: Superiority; p = 0.893, Chi-squared — P-value was based on likelihood ratio chi-square test
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with extreme ovarian responses: AMH >= 15 pmol/L (>=15 oocytes retrieved); Test type: Superiority; p = 0.002, Chi-squared — P-value was based on likelihood ratio chi-square test
Statistical Analysis 3: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with extreme ovarian responses: AMH >= 15 pmol/L (>=20 oocytes retrieved); Test type: Superiority; p = 0.021, Chi-squared — P-value based on likelihood ratio chi-square test

10. Secondary Outcome: Proportion of Participants With Preventive Interventions for Early Ovarian Hyperstimulation Syndrome (OHSS)
Time Frame: ≤9 days after triggering of final follicular maturation
Population: The FAS comprised of all participants randomized or exposed.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants
  Cycle cancellation | 0 | 1.1
  Triggering with GnRH agonist | 1.2 | 1.1
  Administration of dopamine agonist | 0.6 | 1.7

11. Secondary Outcome: Proportions of Participants With Early OHSS (Including OHSS of Moderate/Severe Grade) and/or Preventive Interventions for Early OHSS
Description: Defined as proportion of participants with early OHSS, early OHSS of moderate or severe grade, preventive interventions for early OHSS, early OHSS and/or preventive interventions for early OHSS, and early OHSS of moderate or severe grade and/or preventive interventions for early OHSS are presented.
Time Frame: Up to 9 days after triggering of final follicular maturation
Population: The FAS comprised of all participants randomized and exposed.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants
  Early OHSS (any grade) | 10.0 | 18.6
  Early OHSS (moderate/severe) | 6.5 | 13.0
  Early OHSS (any grade) and/or preventive | 10.6 | 20.9
  Early OHSS (moderate/severe) and/or preventive | 7.6 | 16.4
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportions of participants with early OHSS (any grade); Test type: Superiority; p = 0.017, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with early OHSS (moderate/severe); Test type: Superiority; p = 0.035, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 3: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with early OHSS (any grade) and/or preventive interventions; Test type: Superiority; p = 0.006, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 4: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportion of participants with early OHSS (moderate/severe) and/or preventive interventions; Test type: Superiority; p = 0.009, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors

12. Secondary Outcome: Proportions of Participants With Late OHSS (Including OHSS of Moderate/Severe Grade)
Description: Defined as proportions of participants with late OHSS (including OHSS of moderate/severe grade).
  Late OHSS was defined as OHSS with onset >9 days after triggering of final follicular maturation. The proportion of participants with late OHSS, and late OHSS of moderate or severe grade are presented. All OHSS cases were graded as mild, moderate, or severe.
Time Frame: >9 days after triggering of final follicular maturation
Population: The FAS comprised of all participants randomized or exposed.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants
  Late OHSS (any grade) | 1.2 | 1.1
  Late OHSS (moderate/severe) | 0.6 | 1.1
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportions of participants with late OHSS (any grade); Test type: Superiority; p = 0.968, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Proportions of participants with late OHSS (moderate/severe); Test type: Superiority; p = 0.582, Regression, Logistic — P-value was based on likelihood ratio chi-square test; The model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors

13. Secondary Outcome: Number of Follicles on Stimulation Day 6
Description: Defined as the number of follicles observed in both ovaries at the last transvaginal ultrasound (TVUS) in the stimulation phase (on stimulation Day 6).
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized or exposed participants.
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Follicles | 12.8 (7.2) | 13.3 (7.1)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of follicles on stimulation Day 6 was analyzed; Test type: Superiority; p = 0.198, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

14. Secondary Outcome: Number of Follicles at End-of-stimulation
Description: Defined as the number of follicles observed in both ovaries at the last TVUS in the stimulation phase (end-of-stimulation).
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized or exposed participants.
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Follicles | 14.9 (8.0) | 16.3 (8.8)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of follicles at end-of-stimulation was analyzed; Test type: Superiority; p = 0.036, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

15. Secondary Outcome: Size of Follicles on Stimulation Day 6
Description: Defined as size characteristics of follicles on stimulation Day 6.
  Average size of 3 largest follicles has been presented in this endpoint.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
mm | 12.7 (2.1) | 12.8 (2.0)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The average size of 3 largest follicles was analyzed; Test type: Superiority; p = 0.592, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

16. Secondary Outcome: Size of Follicles at End-of-Stimulation
Description: Defined as size characteristics of follicles at end-of-stimulation.
  Average size of 3 largest follicles has been presented in this endpoint.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
mm | 19.2 (1.5) | 19.4 (1.6)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The average size of 3 largest follicles was analyzed; Test type: Superiority; p = 0.286, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

17. Secondary Outcome: Fertilization Rate
Description: The fertilization rate was defined as the number of oocytes with 2 pronuclei divided by the number of oocytes retrieved.
Time Frame: Day 1 after oocyte retrieval (up to approximately 22 days after start of stimulation)
Population: The FAS comprised all randomized and exposed participants
Measure: Mean (Standard Deviation); unit: percentage of fertilized oocytes
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of fertilized oocytes | 54.5 (26.1) | 57.1 (23.4)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The fertilization rate (number of oocytes with 2 pronuclei divided by the number of oocytes retrieved) was analyzed; Test type: Superiority; p = 0.395, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

18. Secondary Outcome: Number and Quality of Embryos
Description: Number of embryos (total and good-quality) on Day 3 are presented. A good-quality embryo was defined as an embryo with ≥6 blastomeres and fragmentation ≤20% on Day 3.
Time Frame: Day 3 after oocyte retrieval (up to approximately 24 days after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: Embryo
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Embryo
  Number of embryo | 5.8 (4.2) | 7.0 (4.3)
  Number of good-quality embryo | 3.9 (3.3) | 4.6 (3.3)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of embryos on Day 3 was analyzed; Test type: Superiority; p = 0.001, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of good-quality embryos on Day 3 was analyzed; Test type: Superiority; p = 0.004, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

19. Secondary Outcome: Number and Quality of Blastocysts
Description: Number of embryos (total and good-quality) on Day 5 are presented. The quality evaluation of blastocysts consisted of assessment of three parameters, as per the Gardner & Schoolcraft system: blastocyst expansion and hatching status (graded: 1-6), inner cell mass (graded: A-D) and trophectoderm (graded: A-D). A good-quality blastocyst was defined as a blastocyst of grade 3BB or higher.
Time Frame: Day 5 after oocyte retrieval (up to approximately 26 days after start of stimulation)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: Blastocysts
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Blastocysts
  Number of blastocysts | 3.1 (2.7) | 4.2 (3.4)
  Number of good-quality blastocysts | 2.3 (2.3) | 3.0 (2.6)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of blastocysts on Day 5 was analyzed; Test type: Superiority; p < .001, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of good-quality blastocysts on Day 5 was analyzed; Test type: Superiority; p < 0.001, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

20. Secondary Outcome: Circulating Levels of Endocrine Parameters (Follicle-stimulating Hormone [FSH], Luteinising Hormone [LH]) on Stimulation Day 6
Description: The median and inter-quartile range (IQR) of FSH and LH levels on stimulation Day 6 are presented.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 166 | 175
IU/L
  FSH | 15.4 [12.0 to 19.6] | 14.7 [12.8 to 17.3]
  LH | 2.6 [1.5 to 6.2] | 2.8 [1.6 to 5.9]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of FSH on stimulation Day 6; Test type: Superiority; p = 0.228, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; The ANCOVA model included treatment and AMH stratum (<15 pmol/L and ≥15 pmol/L) as fixed factors and log-baseline as covariate; Mean ratio = 1.03, 95% CI 2-sided [0.98 to 1.09] — Mean ratio is equal to FE 999049/FOLLISTIM
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of LH on stimulation Day 6; Test type: Superiority; p = 0.777, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.97, 95% CI 2-sided [0.81 to 1.17] — Mean ratio is equal to FE 999049/FOLLISTIM

21. Secondary Outcome: Circulating Levels of Endocrine Parameters (Follicle-stimulating Hormone [FSH], Luteinising Hormone [LH]) at End-of-stimulation
Description: The median and IQR of FSH and LH levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 172
IU/L
  FSH | 14.3 [11.6 to 19.7] | 16.4 [13.5 to 20.4]
  LH | 1.6 [1.0 to 2.5] | 1.4 [0.9 to 2.3]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of FSH at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.89, 95% CI 2-sided [0.84 to 0.94] — Mean ratio is equal to FE 999049/FOLLISTIM
Statistical Analysis 2: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of LH at end-of-stimulation; Test type: Superiority; p = 0.057, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 1.17, 95% CI 2-sided [1.00 to 1.39] — Mean ratio is equal to FE 999049/FOLLISTIM

22. Secondary Outcome: Circulating Levels of Endocrine Parameter (Estradiol) on Stimulation Day 6
Description: The median and IQR of estradiol levels on stimulation Day 6 are presented.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 166 | 175
pmol/L | 2277.1 [1479.4 to 3580.1] | 2680.0 [1608.8 to 4685.9]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of estradiol on stimulation Day 6; Test type: Superiority; p = 0.002, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.81, 95% CI 2-sided [0.71 to 0.93] — Mean ratio is equal to FE 999049/FOLLISTIM

23. Secondary Outcome: Circulating Levels of Endocrine Parameter (Estradiol) at End-of-stimulation
Description: The median and IQR of estradiol levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 172
pmol/L | 6517.0 [4465.3 to 9033.4] | 7438.8 [5363.6 to 10283.1]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of estradiol at end-of-stimulation; Test type: Superiority; p = 0.003, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.85, 95% CI 2-sided [0.76 to 0.95] — Mean ratio is equal to FE 999049/FOLLISTIM

24. Secondary Outcome: Circulating Levels of Endocrine Parameter (Progesterone) on Stimulation Day 6
Description: The median and IQR of progesterone levels on stimulation Day 6 are presented.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 166 | 175
nmol/L | 1.7 [0.8 to 2.4] | 1.7 [0.8 to 2.65]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of progesterone on stimulation Day 6; Test type: Superiority; p = 0.814, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 1.02, 95% CI 2-sided [0.89 to 1.16] — Mean ratio is equal to FE 999049/FOLLISTIM

25. Secondary Outcome: Circulating Levels of Endocrine Parameter (Progesterone) at End-of-stimulation
Description: The median and IQR of progesterone levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 168 | 172
nmol/L | 2.5 [1.9 to 3.5] | 3.1 [2.3 to 4.3]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of progesterone levels at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.78, 95% CI 2-sided [0.68 to 0.88] — Mean ratio is equal to FE 999049/FOLLISTIM

26. Secondary Outcome: Circulating Levels of Endocrine Parameters (Inhibin A) on Stimulation Day 6
Description: The median and IQR of Inhibin A levels on stimulation Day 6 are presented.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 166 | 175
ng/L | 113.1 [75.1 to 171.9] | 129.8 [81.6 to 210.6]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of Inhibin A on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.82, 95% CI 2-sided [0.73 to 0.92] — Mean ratio is equal to FE 999049/FOLLISTIM

27. Secondary Outcome: Circulating Levels of Endocrine Parameters (Inhibin A) at End-of-stimulation
Description: The median and IQR of Inhibin A levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 172
ng/L | 323.8 [222.1 to 458.8] | 390.3 [301.0 to 551.1]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of Inhibin A at end-of-stimulation; Test type: Superiority; p < 0.001, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.80, 95% CI 2-sided [0.72 to 0.88] — Mean ratio is equal to FE 999049/FOLLISTIM

28. Secondary Outcome: Circulating Levels of Endocrine Parameters (Inhibin B) on Stimulation Day 6
Description: The median and IQR of inhibin B levels on stimulation Day 6 are presented.
Time Frame: At Day 6 of stimulation
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 166 | 175
ng/L | 570.5 [396.0 to 853.0] | 686.0 [431.0 to 1004.0]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of Inhibin B on stimulation Day 6; Test type: Superiority; p < 0.001, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.83, 95% CI 2-sided [0.75 to 0.93] — Mean ratio is equal to FE 999049/FOLLISTIM

29. Secondary Outcome: Circulating Levels of Endocrine Parameters (Inhibin B) at End-of-stimulation
Description: The median and IQR of inhibin B levels at end-of-stimulation are presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The FAS comprised of all randomized and exposed participants.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 169 | 172
ng/L | 686.0 [461.0 to 1057.0] | 734.5 [492.5 to 1120.5]
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); Circulating levels of Inhibin B at end-of-stimulation; Test type: Superiority; p = 0.027, ANCOVA — The P-value corresponds to the two-sided F-test of treatment effect; [statistical method as in outcome 20, analysis 1]; Mean ratio = 0.88, 95% CI 2-sided [0.79 to 0.99] — Mean ratio is equal to FE 999049/FOLLISTIM

30. Secondary Outcome: Number of Stimulation Days
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Days | 8.9 (1.9) | 8.8 (1.7)
Statistical Analysis 1: Comparison: FE 999049 (Follitropin Delta) vs FOLLISTIM (Follitropin Beta); The number of stimulation days at end-of-stimulation; Test type: Superiority; p = 0.694, van Elteren test — 2-sided; P-value was based on van Elteren test adjusted for AMH strata

31. Secondary Outcome: Total Gonadotropin Dose of FE 999049
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | FE 999049 (Follitropin Delta)
Number analyzed (Participants) | 170
μg | 83.5 (28.9)

32. Secondary Outcome: Total Gonadotropin Dose of FOLLISTIM
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 177
IU | 1499 (514)

33. Secondary Outcome: Number of Participants With Adverse Events (AEs) Stratified by Intensity
Description: The frequency of participants with total AEs and AEs by categories of intensity (mild, moderate, severe) are presented. An AE was any untoward medical occurrence in a participants participating in clinical trial. The intensity of AE was classified using the following 3-point scale: mild = awareness of signs or symptoms, but no disruption of usual activity); moderate = event sufficient to affect usual activity (disturbing); or severe = inability to work or perform usual activities (unacceptable).
Time Frame: From signed informed consent up to 5-6 weeks after transfer
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: Participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
Participants
  Any AE | 73 | 92
  Mild AE | 69 | 86
  Moderate AE | 8 | 12
  Severe AE | 0 | 1

34. Secondary Outcome: Proportion of Participants Who Had Markedly Abnormal Value Changes From Baseline in Clinical Chemistry Parameters at End-of-stimulation
Description: Defined as number of participants with at least one markedly abnormal finding in clinical chemistry parameters (as assessed by investigator) were reported. The clinical chemistry parameters included: alanine transaminase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), bicarbonate, bilirubin direct, bilirubin total, blood urea nitrogen, calcium, chloride, cholesterol total, creatinine, gamma-glutamyl transpeptidase, glucose, lactate dehydrogenase, phosphorus, potassium, sodium, total protein, uric acid.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
participants
  ALT (IU/L): Normal to markedly high (>3xULN) | 0 | 1
  AST (IU/L): Normal to markedly high (>3xULN) | 0 | 1

35. Secondary Outcome: Proportion of Participants Who Had Markedly Abnormal Value Changes From Baseline in Hematology Parameters at End-of-stimulation
Description: Defined as number of participants with at least one markedly abnormal changes in hematology parameters (as assessed by investigator) were reported. Hematology parameters included: red blood cells, white blood cells, red blood cells morphology, white blood cells morphology, haemoglobin, haematocrit, mean corpuscular volume, mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, platelets.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
participants | 0 | 0

36. Secondary Outcome: Proportion of Participants Who Had Markedly Abnormal Value Changes From Baseline in Clinical Chemistry Parameters at End-of-trial
Description: as for outcome 34
Time Frame: Up to 5-6 weeks after transfer
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
participants | 0 | 0

37. Secondary Outcome: Proportion of Participants Who Had Markedly Abnormal Value Changes From Baseline in Hematology Parameters at End-of-trial
Description: as for outcome 35
Time Frame: Up to 5-6 weeks after transfer
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
participants
  Leukocytes (10^9/L) Normal to markedly high (>=16) | 0 | 1
  Hemoglobin (g/L) Normal to markedly low | 0 | 1
  Hematocrit (ratio) Normal to markedly low (>=0.56) | 0 | 1

38. Secondary Outcome: Frequency and Intensity of Injection Site Reactions
Description: The presence of of injection site reactions (redness, itching, pain, swelling and bruising) immediately, 30 minutes and 24 hours after the injection are presented. The injection site reactions were assessed as none, mild, moderate and severe. The number of injection site reactions (mild, moderate or severe) based on all assessments performed is presented.
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: events
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
events
  Any mild injection site reaction | 271 | 719
  Any moderate injection site reaction | 7 | 19
  Any severe injection site reaction | 1 | 0
  Mild redness | 140 | 174
  Moderate redness | 2 | 0
  Severe redness | 0 | 0
  Mild itching | 4 | 5
  Moderate itching | 1 | 0
  Severe itching | 0 | 0
  Mild pain | 19 | 411
  Moderate pain | 1 | 16
  Severe pain | 0 | 0
  Mild swelling | 6 | 10
  Moderate swelling | 0 | 0
  Severe swelling | 0 | 0
  Mild bruising | 102 | 119
  Moderate bruising | 3 | 3
  Severe bruising | 1 | 0

39. Secondary Outcome: Technical Malfunctions of the Administration Pens
Time Frame: End-of-stimulation (up to 20 stimulation days)
Population: The safety analysis set comprised of all randomized and exposed participants.
Measure: Number; unit: percentage of participants
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
Number analyzed (Participants) | 170 | 177
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of obtaining informed consent until the last visit (end-of-trial) (up to approximately 2 years) .
Description: Adverse events with onset after start of first administration of IMP were considered treatment -emergent and are presented for the safety analysis set.
Arm/Group | FE 999049 (Follitropin Delta) | FOLLISTIM (Follitropin Beta)
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/177
Serious Adverse Events (participants affected / at risk) | 0/170 | 2/177
Other Adverse Events (participants affected / at risk) | 73/170 | 92/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (Follitropin Delta) (N=170) | FOLLISTIM (Follitropin Beta) (N=177)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (Follitropin Delta) (N=170) | FOLLISTIM (Follitropin Beta) (N=177)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (6)
Injection site erythema (General disorders) | 13 (14) | 15 (15)
Injection site pruritus (General disorders) | 0 (0) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 10 (10)
Abortion spontenous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 19 (19) | 35 (35)
Ovarian cyst (Reproductive system and breast disorders) | 5 (5) | 7 (7)
Ovarian enlargement (Reproductive system and breast disorders) | 5 (5) | 5 (5)
Pelvic fluid collection (Reproductive system and breast disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03228680/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT03228680/SAP_001.pdf